CLINICAL TRIAL: NCT04033003
Title: Group Antenatal Care to Promote a Healthy Pregnancy and Optimize Maternal and Newborn Outcomes: A Cluster Randomized Controlled Trial
Brief Title: Group Antenatal Care and Delivery Project
Acronym: GRAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Dodowa Health Research Centre (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jody Rae Lori, Professor & Associate Dean for Global Affairs, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00161464; R01HD096277 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-07-25 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Antenatal Care
Keywords: Antenatal care; Sub-Saharan Africa; Ghana

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ANC (Experimental): Intervention groups consist of up to 14 women of similar gestation age (10 to 20 weeks) for nine meetings. The first meeting is an individual meeting with the midwife and the standard history and physical exam as well as lab tests are completed. Group meetings are held once a month until 28 weeks of pregnancy, then every 2 weeks until 34 weeks of pregnancy, and the remaining group meetings are once a week. Prior to the start of each group, blood pressure, weight, and a urinalysis are measured for each woman.
  Interventions: Behavioral: Group ANC
- Stand ANC (No Intervention): Individual standard antenatal care delivered at health facilities in Ghana

INTERVENTIONS:
Behavioral: Group ANC — Intervention groups of up to 14 women of similar gestation age (10 to 20 weeks) for nine meetings. The first meeting is an individual meeting with the midwife and the standard history and physical exam as well as lab tests are completed. Group meetings are held once a month until 28 weeks of pregnancy, then every 2 weeks until 34 weeks of pregnancy, and the remaining group meetings are once a week. Prior to the start of each group, blood pressure, weight, and a urinalysis are measured for each woman.
  Arms: Group ANC

SUMMARY:
Antenatal care (ANC) has the potential to play a pivotal role in ensuring positive pregnancy outcomes for both mothers and their newborns. A critical component of all ANC is teaching women to recognize the major complications that account for the majority of preventable maternal and newborn deaths. Antenatal care provides an opportunity to promote a healthy lifestyle, to integrate positive health behaviors, and to develop a trusting relationship with a provider and the health system. While group ANC has been delivered and studied in high-resource settings for over a decade, it has only recently been introduced as an alternative to individual care in sub-Saharan Africa.

The goal of this research is to improve health literacy and reduce preventable maternal and newborn morbidities and mortality within highly vulnerable, low and non-literate populations that assume a disproportionate burden of poor pregnancy outcomes globally. This research examines a bold, new approach to ANC that takes provision of care out of clinic exam rooms into small groups of women grouped by gestational age in low resource settings with low and non-literate populations. Group ANC has the potential to shift the current clinical practice paradigm of antenatal care for highly vulnerable women to improve maternal and newborn outcomes both globally and domestically.

The investigators hypothesize that pregnant women randomized into group ANC will exhibit increased health literacy through: 1) increased birth preparedness and complication readiness (BPCR), including recognition of danger signs and knowledge of how to respond to such signs; 2) higher rates of care-seeking behaviors, including seeking care for problems identified during pregnancy, higher facility delivery rates, and increased attendance at postnatal and postpartum care; and 3) better clinical outcomes for themselves and their newborns than women who received the routine, individual ANC.

DETAILED DESCRIPTION:
We are at a critical time to examine new, innovative strategies to promote healthy pregnancy and optimize maternal and newborn outcomes. Generating successful strategies will require careful examination of existing service delivery models, challenging the current structure of care provision. One aspect of care, recently identified by the World Health Organization, which merits further research, is group antenatal care (ANC).

Since ANC is widely available and attended by the majority of pregnant women in Ghana without the expected impact on birth outcomes, it is vital to examine the way antenatal health messages are delivered. Pregnant women must receive health information that is accurate and easy to understand for them to make informed choices to improve their health and the health of their baby. A critical component of all ANC is teaching women to recognize the major complications that account for the majority of preventable maternal and newborn deaths. Antenatal care provides an opportunity to promote a healthy lifestyle, to integrate positive health behaviors, and to develop a trusting relationship with a provider and the health system. Interactions during ANC provide the opportunity to identify and treat numerous problems, as well as providing a setting to improve women's health literacy. Patients must receive health messages in a manner that allows them to process and evaluate the information and ultimately use it to impact their own health.

The effectiveness of ANC depends on the multidimensional concept of health literacy. Initially considered only as a patient's ability to read and understand written information, it is now more broadly defined as a person's ability to acquire or access information, understand it, and use the information in ways that promote and maintain good health. Despite a burgeoning emphasis on health literacy in high resource countries, there are a dearth of studies examining interventions to improve health literacy in low-resource settings. Even fewer studies have examined maternal health literacy, defined as the "cognitive and social skills which determine the motivation and ability of women to gain access to, understand, and use information in ways that promote and maintain their health and that of their children''. New approaches to improve health literacy are sorely needed in countries where women and newborns continue to die from preventable causes.

Antenatal care has been delivered the same way for decades. Clinics and hospitals in low-resource countries are notorious for providing ethnocentric care, privileging northern medical values at the expense of traditional and community values. Yet health literacy is affected by the cultural context in which learning takes place, including, but not limited to, belief systems, traditions, understanding, and communication styles. Transmitting health information in a clinical setting often fails to take into account the social and economic circumstances of patients, therefore not achieving the expected impact on health behaviors. This divide has contributed to a lack of progress in reaching the most vulnerable populations. If pregnant women do not receive health messages in a comprehensible way, they cannot effectively maximize the benefits of the health system. Substantially improving women's ability to understand and utilize health information is of utmost importance if we are to reach the global targets of 70 maternal deaths per 100,000 live births by 2030 and a neonatal mortality rate of 12 per 1000 live births set by WHO/USAID.

The investigators hypothesize that pregnant women randomized into group ANC will exhibit increased health literacy through:

1. Increased BPCR, including recognition of danger signs and knowledge of how to respond to such signs
2. Higher rates of care-seeking behaviors, including seeking care for problems identified during pregnancy, higher facility delivery rates, and increased attendance at postnatal and postpartum care
3. Better clinical outcomes for themselves and their newborns than women who received the routine, individual ANC.

The intervention consists of nine meetings; one individual meeting and eight group meetings. At the initial ANC visit, women are assigned to a small groups with up to14 women of similar gestational age. Women meet individually with the midwife and the standard history and physical exam as well as lab tests are completed; group visits start at the second ANC visit. Prior to the start of each group, blood pressure, weight, and a urinalysis are measured for each woman. The midwife, health facility staff member, and patients then sit in circle facing one another for a 60-90 minute facilitated discussion. The health facility staff member will assist the midwife with group activities. The model uses strategies such as story-telling, peer support, and demonstration and teach-back to enhance its effectiveness. Health literacy is incorporated as an integral part of clinical practice within the model - not as an add-on to care.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the study
* less than 20 weeks' gestation 3) able to speak Dangme, Ga, Akan, Ewe, or English
* over the age of 15 years

Exclusion Criteria:

* No history of medical problems that would indicate the participant might be considered "high risk" (e.g., hypertension, insulin-dependent diabetes mellitus) and thus requiring a more individualized approach to care.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Study for pregnant women
Enrollment: 1761 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John EO Williams, Study Director — Dodowa Health Research Centre; Jody R Lori, PhD, Principal Investigator — University of Michigan
Locations (14):
- Ghana (14):
  - Adawso Health Center, Adawso
  - Adukrom Health Center, Adukrom
  - Klo Agogo Polyclinic, Agogo
  - Abiriw Clinic, Akropong
  - St Martin's Hospital, Akropong
  - Akuse Hospital, Akuse
  - Nkurakan Health Center, Koforidua
  - Tetteh Quarshie Hospital, Mampong
  - Adoagyiri Health Center, Nsawam
  - Djankrom Health Center, Nsawam
  - Nsawam Health Center, Nsawam
  - Nsawam Hospital, Nsawam
  - Atua Hospital, Somanya
  - Somanya Polyclinic, Somanya

REFERENCES:
- [Derived] Lanyo TN, Williams JEO, Ghosh B, Apetorgbor VEA, Kukula VA, Zielinski R, Awini E, Moyer CA, Lori J. Impact of group antenatal care on lactational amenorrhea method awareness and knowledge: A cluster randomized control trial. PLoS One. 2025 Oct 15;20(10):e0333074. doi: 10.1371/journal.pone.0333074. eCollection 2025. PMID 41091707
- [Derived] Apetorgbor V, Awini E, Ghosh B, Zielinski R, Amankwah G, Kukula VA, James K, Williams JEO, Lori JR, Moyer CA. The impact of group antenatal care on newborns: Results of a cluster randomized control trial in Eastern Region, Ghana. BMC Pediatr. 2024 Nov 18;24(1):747. doi: 10.1186/s12887-024-05225-9. PMID 39558280
- [Derived] Kukula VA, Awini E, Ghosh B, Apetorgbor V, Zielinski R, Amankwah G, Ofosu WK, James K, Williams JEO, Lori JR, Moyer CA. Effect of group antenatal care versus individualized antenatal care on birth preparedness and complication readiness: a cluster randomized controlled study among pregnant women in Eastern Region of Ghana. BMC Pregnancy Childbirth. 2024 Aug 16;24(1):546. doi: 10.1186/s12884-024-06743-1. PMID 39152408
- [Derived] Lori JR, Williams JEO, Kukula VA, Apetorgbor VEA, Awini EA, Amankwah G, Zielinski R, Lockhart N, James KH, Moyer CA. Group Antenatal Care in Ghana: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2022 Sep 9;11(9):e40828. doi: 10.2196/40828. PMID 36083608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourteen health facilities were randomized using a matched-pair method. Variables for matching included the number of deliveries and the average gestational age of pregnancy at the time of enrollment, so that facilities within each pair are similar to each other. For each pair of facilities, one site was randomly assigned to group ANC (intervention) and the other to routine individual ANC (control). Individual women were recruited at each health facility.
Units Other Than Participants: Health Facilities
Period: T0 (Baseline at Recruitment)
Arm/Group | Group ANC | Stand ANC
Started | 877; 7 Health Facilities | 884; 7 Health Facilities
Completed | 877; 7 Health Facilities | 884; 7 Health Facilities
Not Completed | 0; 0 Health Facilities | 0; 0 Health Facilities
Period: T1 (34 Wks Gestation - 3 Wks Postpartum)
Arm/Group | Group ANC | Stand ANC
Started | 877; 7 Health Facilities | 884; 7 Health Facilities
Completed | 617; 7 Health Facilities | 668; 7 Health Facilities
Not Completed | 260; 0 Health Facilities | 216; 0 Health Facilities
Not completed — Lost to Follow-up | 113 | 190
Not completed — Protocol Violation | 115 | 0
Not completed — Withdrawal by Subject | 2 | 6
Not completed — No longer meets criteria | 30 | 19
Not completed — Death | 0 | 1
Period: T2 (6 - 12 Weeks Postpartum)
Arm/Group | Group ANC | Stand ANC
Started | 730; 7 Health Facilities (The participants lost-to-follow up in T1 (third trimester) are eligible to participate in T2 (post-delivery) survey, which is why the number of participants started in T2 does not equal those who completed T1. The number started T2 is the sum of T1 completed + T1 lost-to-follow-up.) | 858; 7 Health Facilities (The participants lost-to-follow up in T1 (third trimester) are eligible to participate in T2 (post-delivery) survey, which is why the number of participants started in T2 does not equal those who completed T1. The number started T2 is the sum of T1 completed + T1 lost-to-follow-up.)
Completed | 585; 7 Health Facilities | 596; 7 Health Facilities
Not Completed | 145; 0 Health Facilities | 262; 0 Health Facilities
Not completed — Lost to Follow-up | 133 | 247
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — No longer meets criteria | 1 | 10
Not completed — Death | 2 | 2
Period: T3 (5 - 8 Month Postpartum)
Arm/Group | Group ANC | Stand ANC
Started (The participants lost-to-follow up in T 2 are eligible to participate in T3 survey, which is why the number of participants started in T3 does not equal those who completed T2. The number started T3 is the sum of T2 completed + T2 lost-to-follow-up.) | 718; 7 Health Facilities | 843; 7 Health Facilities
Completed | 619; 7 Health Facilities | 673; 7 Health Facilities
Not Completed | 99; 0 Health Facilities | 170; 0 Health Facilities
Not completed — Lost to Follow-up | 96 | 165
Not completed — Withdrawal by Subject | 3 | 5
Period: T4 (11 -14 Months Postpartum)
Arm/Group | Group ANC | Stand ANC
Started (The participants lost-to-follow up in T3 are eligible to participate in T4 survey, which is why the number of participants started in T4 does not equal those who completed T3. The number started T4 is the sum of T3 completed + T3 lost-to-follow-up.) | 715; 7 Health Facilities | 838; 7 Health Facilities
Completed | 626; 7 Health Facilities | 688; 7 Health Facilities
Not Completed | 89; 0 Health Facilities | 150; 0 Health Facilities
Not completed — Lost to Follow-up | 89 | 150

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group ANC | Stand ANC | Total
Number analyzed (Participants) | 877 | 884 | 1761
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 40 | 69
  Between 18 and 65 years | 848 | 844 | 1692
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 877 | 884 | 1761
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Ghana | 877 | 884 | 1761

OUTCOME MEASURES:

1. Primary Outcome: Change in Ability to Identify Danger Signs in Pregnancy
Description: Ability to identify danger signs in pregnancy will be measured utilizing a self-report, open ended, question that asks participants to identify warning signs that may occur during pregnancy (e.g. headache, vision changes, fever, vaginal bleeding, swollen face, etc.). There is no validated or standardized instrument to measure Birth Preparedness and Complication Readiness (BPCR).
  The measure used in this study is an open-end question: What are the danger signs during pregnancy? Things that might mean there is a problem with you or the baby. Fourteen possible correct responses; raw item scores are a sum of individual responses; scores range from 0 to 14. Reported results are the average of all individual scores within the study arm. Change will be measured by calculating the difference in the mean at T0 and T1. Higher score means a better outcome.
Time Frame: T0 Baseline (at recruitment) and T1 (34 weeks gestation - 3 weeks postdelivery)
Population: Group ANC: Number of participants analyzed at T0 = 877; Number of participants analyzed at T1 = 617 Standard ANC: Number of participants analyzed at T0 = 884; Number of participants analyzed at T1 = 668
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 877 | 884
units on a scale
  T0 - baseline | 1.8 (1.3) | 1.7 (1.4)
  T1 (34 weeks gestation - 3 weeks postdelivery): number analyzed (Participants) | 617 | 688
  T1 (34 weeks gestation - 3 weeks postdelivery) | 3.4 (1.6) | 2.2 (1.3)

2. Primary Outcome: Change in Birth Preparedness and Complication Readiness
Description: Change in the ability to identify a strategy for birth preparedness and complication readiness (BPCR) will be measured using a binary response (yes/no) to a question that ask participants if they have: (1) saved money, (2) identified birth facility for delivery, (3) identified emergency transportation to the facility, and (4) identified a blood donor. There is no validated or standardized instrument to measure BPCR. The measure used in this study is an open-end question: What are some things a woman can do to prepare for birth? Eleven possible correct responses; raw item scores are a sum of individual responses; scores range from 0 to 11. Reported results are the average of all individual scores within the study arm. Change will be measured by calculating the difference in the mean at T0 and T1. Higher score means a better outcome.
Time Frame: T0 (Baseline at recruitment) and T1 (34 weeks gestation - 3 weeks postdelivery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 877 | 884
units on a scale
  T0 | 1.4 (0.9) | 1.42 (0.9)
  T1 (34 weeks gestation - 3 weeks postdelivery): number analyzed (Participants) | 617 | 668
  T1 (34 weeks gestation - 3 weeks postdelivery) | 2.9 (1.5) | 1.7 (1.0)

3. Primary Outcome: Change in Ability to Identify Newborn Danger Signs
Description: Ability to identify newborn danger signs will be measured utilizing a self-report, open ended, question that asks participants to identify newborn danger signs that may occur after delivery (e.g. poor suck, jaundice, difficulty/fast breathing, and convulsions). Change will be measured by calculating the difference in the mean at T0 and T1.
  There is no validated or standardized instrument to measure Birth Preparedness and Complication Readiness (BPCR). The measure used in this study is an open-end question: What are the danger signs for your newborn? Things that might mean there is a problem. Thirteen possible correct responses; raw item scores are a sum of individual responses; scores range from 0 to 13. Reported results are the average of all individual scores within the study arm. Higher score means a better outcome.
Time Frame: T0 (Baseline at recruitment) and T1 (34 weeks gestation - 3 weeks postdelivery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 877 | 884
units on a scale
  T0 Baseline at recruitment | 1.9 (1.2) | 1.5 (1.2)
  T1 (34 weeks gestation - 3 weeks postdelivery): number analyzed (Participants) | 617 | 668
  T1 (34 weeks gestation - 3 weeks postdelivery) | 1.8 (1.3) | 2.8 (1.5)

4. Primary Outcome: Attendance of ANC Visits
Description: Attendance of 4 or more ANC visits will be gleaned from data reported on the participant's ANC/health card.
Time Frame: T2 (6-12 weeks after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 557 | 526
Participants
  Yes | 555 | 523
  No | 2 | 3

5. Primary Outcome: Place of Delivery
Description: Place of delivery will be measured using a self-report question (facility delivery, home delivery).
Time Frame: T2 (6-12 weeks after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 585 | 593
Participants
  Delivered at health facility | 567 | 567
  Delivered at home | 18 | 26

6. Primary Outcome: Attendance at Postpartum Check-ups for Mother
Description: Attendance of postpartum check-ups will be gleaned from information on the participant's ANC/health card.
Time Frame: T2 (6-12 weeks after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 584 | 591
Participants
  Attended 2 day pp visit | 392 | 451
  Attended 6 day pp visit | 469 | 447
  Attended 6 week pp visit | 517 | 541

7. Primary Outcome: Attendance at Postnatal Check-up for Newborn
Description: Attendance of postnatal checkup will be gleaned from information on the participant's ANC/health card using a measure of 3 visits before 6 weeks for newborns.
Time Frame: T2 (6-12 weeks after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 580 | 585
Participants
  2 day postnatal visit | 412 | 460
  6 day postnatal visit | 473 | 453
  6 week postnatal visit | 531 | 550

8. Primary Outcome: Birth Outcome
Description: Birth outcomes will be self-reported and measured as stillbirth, live birth, early neonatal mortality.
Time Frame: T2 (6-12 weeks after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 585 | 595
Participants
  Live birth | 580 | 587
  Stillbirth | 5 | 8
  Early neonatal mortality | 6 | 7

9. Primary Outcome: Change in Health Literacy
Description: Change in Health Literacy will be measured using the Maternal Health Literacy Scale. Change over time will be analyzed using between group analysis and calculating the difference in the mean from T0 to T2.
  Maternal Health Literacy (MaHeLi) scale is a validated measure that consists of 12 yes-or-no questions to assess maternal health literacy among the participants. Raw item scores are a sum of individual responses; scores range from 0 to 12. Reported results are the average of all individual scores within the study arm. Higher score means a better outcome.
Time Frame: T0 (Baseline at recruitment) and T2 (6 - 12 weeks postdelivery)
Population: Group ANC: Number of participants analyzed at T0 = 877; Number of participants analyzed at T2 = 585 Standard ANC: Number of participants analyzed at T0 = 884; Number of participants analyzed at T2 = 596
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 887 | 884
score on a scale
  T0 - baseline: number analyzed (Participants) | 877 | 884
  T0 - baseline | 9.6 (1.7) | 9.7 (1.6)
  T2 - 6 weeks post-delivery: number analyzed (Participants) | 585 | 596
  T2 - 6 weeks post-delivery | 11.3 (0.9) | 11 (1.2)

10. Secondary Outcome: Change in Ability to Identify Postpartum Danger Signs for Mother
Description: Ability to identify danger signs after delivery will be measured utilizing a self-report, open ended, question that asks participants to identify warning signs that may occur after delivery (e.g. increased bleeding or large clots; weakness/fainting; fever; pain in abdominal or breast; painful urination, etc.). Change will be measured by calculating the difference in the mean at T0 (baseline) and T1 (34 weeks gestation - 3 weeks postdelivery).
  There is no validated or standardized instrument to measure postpartum danger signs. The measure used in this study is an open-end question: What are the danger signs for you, the mother, after the baby is born? Fourteen possible correct responses; raw item scores are a sum of individual responses; scores range from 0 to 14. Reported results are the average of all individual scores within the study arm. Change will be measured by calculating the difference in the mean at T0 and T1. Higher score means a better outcome.
Time Frame: T0 (Baseline at recruitment) and T1 (34 weeks gestation - 3 weeks postdelivery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 877 | 884
units on a scale
  T0 | 1.26 (1.1) | 1.17 (1.1)
  T1: number analyzed (Participants) | 617 | 668
  T1 | 2.44 (1.3) | 1.69 (1.2)

11. Secondary Outcome: Change in Ability to Identify the Recommended Action Steps When a Problem is Identified
Description: Ability of mother to identify recommended action steps in response to danger signs that may occur before or after delivery. There is no validated or standardized instrument to measure this outcome, therefore the measure used in this study is the question: What do you think you would do if you have any of these (danger signs)? Responses are coded as Go to hospital or health facility CHECKED (1) or Go to hospital or health facility NOT CHECKED (0). Reported results are the sum of individual responses; higher score "Go to hospital checked" means a better outcome.
Time Frame: T0 (Baseline at recruitment) and T1 (34 weeks gestation - 3 weeks postdelivery)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 877 | 884
Participants
  T0: Go to hospital or health facility CHECKED | 671 | 636
  T0: Go to hospital or health facility NOT CHECKED | 206 | 248
  T1: number analyzed (Participants) | 617 | 668
  T1: Go to hospital or health facility CHECKED | 594 | 552
  T1: Go to hospital or health facility NOT CHECKED | 23 | 116

12. Secondary Outcome: Change in Knowledge of Family Planning Methods
Description: Knowledge of family planning methods will be measured by self-report using a question that asks participants to identify all the methods of family planning they know. Change will be measured by calculating the difference in the mean at baseline and 3rd trimester.
  There is no validated or standardized instrument to measure this outcome, therefore the measure used in this study is an open-end question that asks participants to identify all the methods of family planning they know. Change will be measured by calculating the difference in the mean at T0 (baseline) and T1 (34 weeks gestation - 3 weeks postdelivery). There are eleven possible correct responses; raw item scores are a sum of individual responses; scores range from 0 to 11. Reported results are the average of all individual scores within the study arm. Change will be measured by calculating the difference in the mean at T0 and T1. Higher score means a better outcome.
Time Frame: T0 (Baseline at recruitment) and T1 (34 weeks gestation - 3 weeks postdelivery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 877 | 884
units on a scale
  T0 | 2.22 (1.3) | 2.01 (1.39)
  T1: number analyzed (Participants) | 617 | 668
  T1 | 3.88 (1.7) | 2.37 (1.4)

13. Secondary Outcome: Change in Intent to Use Family Planning
Description: Intent to use family planning methods will be measured by self-report using a binary (yes/no) question that asks participants, "Do you intend to use family planning after delivery?". Responses are coded as yes = 1 or no = 0. A higher number equals those who indicated yes to their intent to use family planning after delivery. Change over time will be analyzed using between group analysis and calculating the difference in the mean from T0 (baseline) to T1( 34 weeks gestation - 3 weeks postdelivery).
Time Frame: T0 (Baseline at recruitment) and T1 (34 weeks gestation - 3 weeks postdelivery)
Population: Group ANC: Number of participants analyzed at T0 = 747; Number of participants analyzed at T1 = 526 Standard ANC: Number of participants analyzed at T0 = 760; Number of participants analyzed at T1 = 525
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 747 | 760
units on a scale
  T0 | 0.38 (0.5) | 0.41 (0.5)
  T1: number analyzed (Participants) | 526 | 525
  T1 | 0.61 (0.5) | 0.42 (0.5)

14. Secondary Outcome: Change in Uptake of Family Planning
Description: Uptake of family planning will be measured by self-report using a binary (yes/no) question that asks participants if they are currently using any family planning method. Responses are coded as yes = 1 or no = 0. A higher number equals those who indicated "yes" to currently using family planning. Change over time will be analyzed using between group analysis and calculating the difference in the mean from T2 (6-12 weeks after delivery), T3 (5 - 8 months postpartum), and T4 (11 - 14 months postpartum).
Time Frame: T2 (6-12 weeks after delivery), T3 (5 - 8 months postpartum), and T4 (11 - 14 months postpartum)
Population: Group ANC: Number of participants analyzed at T2 = 585; Number analyzed at T3 = 619; Number analyzed at T4 = 609 Standard ANC: Number of participants analyzed at T0 592= ; Number analyzed at T1 = 673; Number analyzed at T4 = 674 Participants lost to follow-up at T2 and T3 remain eligible to complete surveys at subsequent timepoints. Thus, there may be more participants analyzed at later timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 619 | 674
units on a scale
  T2: number analyzed (Participants) | 585 | 592
  T2 | 0.15 (0.4) | 0.09 (0.3)
  T3: number analyzed (Participants) | 619 | 673
  T3 | 0.25 (0.4) | 0.2 (0.4)
  T4: number analyzed (Participants) | 609 | 674
  T4 | 0.35 (0.5) | 0.43 (0.5)

15. Secondary Outcome: Change in Interpersonal Violence
Description: Experiences of physical, sexual, and emotional violence were measured using an investigator-derived questionnaire that asks participants if they experienced violence in the past year, and if resources and support are available to them. Raw item scores are a sum of individual responses; scores range from 0 to 9. Reported results are the average of all individual scores within the study arm. Change will be measured by calculating the difference in the mean at T0 and T4. Higher score means higher rates of reported sexual and emotional violence and lower access to resources and support.
  Change over time will be analyzed using between group analysis and calculating the difference in the mean from T0 (baseline) to T4 (11 - 14 months postpartum)
Time Frame: T0 (baseline) and T4 (11 - 14 months postpartum)
Population: Group ANC: Number of participants analyzed at T0 = 873 ; Number of participants analyzed at T4 = 626 Standard ANC: Number of participants analyzed at T0 = 884; Number of participants analyzed at T4 = 686
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 873 | 884
units on a scale
  T0 | 4.48 (1.4) | 4.59 (1.4)
  T4: number analyzed (Participants) | 626 | 686
  T4 | 4.62 (1.0) | 4.78 (0.8)

16. Secondary Outcome: Experience of ANC Care
Description: Experience of ANC care is measured using a twenty-one item investigator-derived questionnaire that asks participants about their experience regarding respectful care, satisfaction with care, and experience such as privacy and treatment with health system during their ANC visits. Raw item scores are a sum of individual responses; scores range from 0 to 21. Reported results are the average of all individual scores within the study arm. Higher score means a better outcome.
Time Frame: T2 (6-12 postpartum)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 585 | 592
units on a scale | 20.1 (1.4) | 18.79 (2.1)

17. Secondary Outcome: Completion of IPTp2 Malaria Prophylaxis During Pregnancy
Description: Data gleaned from the participant's ANC/health record will be used to measure affirmative completion of IPTp2 malaria prophylaxis during pregnancy.
Time Frame: T1 (34 weeks gestation - 3 weeks postdelivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 612 | 657
Participants
  YES (completed IPTp2 malaria prophylaxis during pregnancy) | 375 | 419
  NO (did not complete IPTp2 malaria prophylaxis during pregnancy) | 237 | 238

18. Secondary Outcome: Completion of Least Two Tetanus Toxoid Vaccines During Pregnancy
Description: Data gleaned from the participant's ANC/health record will be used to measure if the participant received least two tetanus toxoid vaccines during pregnancy.
Time Frame: T1 (34 weeks gestation - 3 weeks postdelivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 611 | 660
Participants
  YES (received at least two tetanus toxoid vaccines during pregnancy) | 487 | 518
  No (did not receive at least two tetanus toxoid vaccines during pregnancy) | 124 | 142

19. Secondary Outcome: Newborn Weight
Description: Newborn weight in grams; these data will be retrieved from the participant's ANC/health card and measured as newborn weight.
Time Frame: T2 (6-12 weeks postpartum)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 492 | 469
Participants
  ≥ 2500 g | 459 | 431
  < 2500 g | 33 | 38

20. Secondary Outcome: Mother's Hemoglobin at Delivery in Grams Per Deciliter (g/dl).
Description: Mother's hemoglobin at delivery; these data will be retrieved from the participant's ANC/health card and measured as hemoglobin in grams per deciliter (g/dl).
Time Frame: T2 (6 - 12 weeks postpartum)
Measure: Count of Participants; unit: Participants
Arm/Group | Group ANC | Stand ANC
Number analyzed (Participants) | 491 | 493
Participants
  Severely anemic (< 7.5) | 4 | 3
  Moderately anemic (> 7.5, <11) | 176 | 177
  Normal (>11) | 311 | 313

ADVERSE EVENTS:
Time Frame: from time of enrollment until study completion (11-14 months post delivery)
Description: clinicaltrials.gov definition
Arm/Group | Group ANC | Stand ANC
All-Cause Mortality (participants affected / at risk) | 2/877 | 3/884
Serious Adverse Events (participants affected / at risk) | 2/877 | 3/884
Other Adverse Events (participants affected / at risk) | 0/877 | 0/884
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group ANC (N=877) | Stand ANC (N=884)
Death not related to study protocol (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) — Death not related to study protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04033003/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04033003/ICF_001.pdf